CLINICAL TRIAL: NCT02145559
Title: A Pharmacodynamic Study of Sirolimus and Metformin in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB13-0614
Record Dates: First submitted 2014-05-19; First posted 2014-05-23 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Breast Neoplasms; Lung Neoplasms; Cancer of Liver; Lymphoma; Cancer of Kidney
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Liver Neoplasms; Lymphoma; Kidney Neoplasms | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin XR (Experimental): All eligible patients with histologically-confirmed advanced solid tumors will be started on sirolimus (3 mg daily) alone for the first 7 days. On day 8, patients will recieve metformin XR (500 mg daily with the evening meal)(through day 21). On day 15, patients randomized to metformin XR will have their dose increased to 1000 mg daily if there is no grade ≥ 2 toxicity due to metformin XR. Patients who develop grade 2 toxicity due to metformin will be maintained on metformin XR 500 mg daily for the rest of the study, while patients who develop > grade 2 toxicity will be taken off study. From day 22 onwards, all patients will be on combination of sirolimus and metformin.
  Interventions: Drug: Metformin XR; Drug: Sirolimus
- Delayed Metformin (Active Comparator): All eligible patients with histologically-confirmed advanced solid tumors will be started on sirolimus (3 mg daily) alone for the first 7 days. On day 8, patients will be randomized to receive no metformin for two weeks (through day 21). From day 22 onwards, all patients will be on combination of sirolimus and metformin. Patients who were initially not randomized to metformin XR will begin taking it at 500 mg daily with an evening meal and titrated up to 1000 mg daily after one week, as above. Each cycle will be 4 weeks.
  Interventions: Drug: Delayed Metformin; Drug: Sirolimus

INTERVENTIONS:
Drug: Metformin XR
  Arms: Metformin XR
Drug: Delayed Metformin
  Arms: Delayed Metformin
Drug: Sirolimus

SUMMARY:
Given the role of mTOR signaling and probable synergistic activity of combining sirolimus and metformin in patients with advanced solid tumors, the investigators hypothesize that:

1. The combination of metformin plus sirolimus will result in reduction of p4EBP1, p70S6K and pAKT more than sirolimus alone in peripheral blood T cells (PBTC).
2. The combination of metformin plus sirolimus will result in decreased levels of serum biomarkers including fasting insulin, C-peptide, glucose, triglycerides, LDH, IGF-1, IGF-1R, IGF-BP and leptin, but an increase in adiponectin in peripheral blood.
3. Expression of active forms of AMPK, mTOR, PI3K, PTEN loss, AKT, LKB1, P62, LC3, and/or ULK1 in the tumor tissue (original pathology) will be predictive of response to combination therapy. This will be an exploratory hypothesis for this study.
4. Sirolimus induced toxicity, especially hyperglycemia and hypertriglyceridemia, will be mitigated by combining sirolimus with metformin.
5. Metformin plus sirolimus will have promising anti-cancer activity and this activity will correlate with decreases in the above biomarkers. This will be an exploratory hypothesis for this study.

DETAILED DESCRIPTION:
Objectives:

This is a descriptive study to evaluate the pharmacodynamic markers of dual sirolimus and metformin therapy.

Primary Objective:

i. To compare the change in the pharmacodynamic biomarker p70S6K in peripheral blood T cells with the combination of metformin XR and sirolimus to that with sirolimus alone.

Secondary Objectives:

i. To compare the changes in pharmacodynamic biomarkers p4EBP1 and pAKT in peripheral blood T cells with the combination of metformin XR and sirolimus to those with sirolimus alone.

ii. To assess the tolerability of the combination of metformin XR plus sirolimus at the selected doses.

iii. To compare fasting serum glucose and triglycerides on sirolimus before and after the addition of metformin XR.

Study Design:

This will be an open-label, randomized study in which all eligible patients with histologically-confirmed advanced solid tumors will be started on sirolimus (3 mg daily) alone for the first 7 days (lead-in period); cycle 1, days 1-8. Before starting the sirolimus the investigators will obtain previous pathology (if available) and collect blood lymphocytes for baseline testing of biomarkers as is shown in study calendar. The pharmacodynamic biomarkers will be collected again on cycle 1, day 8 to assess the effect of sirolimus alone on these biomarkers. In the previous study, the effect of sirolimus on p70S6K was observed within 48 hours of the first dose9. On day 8, patients will be randomized 1:1 to metformin XR (500 mg daily with the evening meal) or no metformin for two weeks (through day 21). On day 15, patients randomized to metformin XR will have their dose increased to 1000 mg daily if there is no grade ≥ 2 toxicity due to metformin XR. Patients who develop grade 2 toxicity due to metformin will be maintained on metformin XR 500 mg daily for the rest of the study, while patients who develop > grade 2 toxicity will be taken off study. A repeat biomarkers evaluation will be done on cycle 1, day 22 to assess the effect of adding metformin on these pharmacodynamic biomarkers. From day 22 onwards, all patients will be on combination of sirolimus and metformin. Patients who were initially not randomized to metformin XR will begin taking it at 500 mg daily with an evening meal and titrated up to 1000 mg daily after one week, as above. Each cycle will be 4 weeks. CT scans will be obtained after every 2 cycles to assess the response by RECIST version 1.140. Metformin will be temporarily held on the day of CT scan and resumed 48 hours after CT scan. This is due to increased risk of lactic acidosis with iodinated contrast agent and is a standard procedure for contrast enhanced CT scan at the University of Chicago.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed solid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
2. ECOG performance status 0 or 1 (See Appendix B).
3. Age ≥ 18 years.
4. Non-pregnant, non-lactating women using adequate contraception.
5. Ability to understand and willingness to sign informed consent.
6. Adequate hematologic, renal and hepatic function, as defined by each of the following:

   * Absolute neutrophil count (ANC) > l500/μl
   * Platelets > 100,000/μl
   * Total bilirubin < 1.5 x upper limit of normal
   * SGOT and SGPT < 2.5x upper limit of normal for patients without liver metastases or SGOT and
   * SGPT < 5 x upper limit of normal for patients with liver metastases.
   * Creatinine < 1.4 mg/dl for females or < 1.5 mg/dl for males.
7. Prior treatment with mTOR inhibitors will be allowed as long as the patient did not have ≥ Grade 3 toxicity attributed to the mTOR inhibitor with prior therapy.
8. Measurable or non-measurable disease will be allowed.
9. Patients taking substrates, inhibitors, or inducers of CYP3A4 (See Appendix C) should be encouraged to switch to alternative drugs whenever possible, given the potential for drug-drug interactions with sirolimus.

Exclusion Criteria

1. Prior treatment with an mTOR inhibitor (including sirolimus) is allowed; however, patients with ≥ grade 3 toxicities with an mTOR inhibitor are excluded.
2. Fasting glucose > 200 mg/dL or fasting triglycerides > 300 mg/dL.
3. Patients who have had chemotherapy or immunotherapy within 4 weeks of starting study drug, or radiotherapy within 14 days of starting study drug, or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
4. Patients may not be receiving any other investigational agents or any concomitant antineoplastic therapy, with the exceptions of octreotide LAR (for neuroendocrine tumors) and endocrine therapy (for prostate, breast, or gynecologic malignancies).
5. Serious underlying medical (including acute decompensated congestive heart failure) or psychiatric illnesses that would, in the opinion of the treating physician, substantially increase the risk for complications related to treatment. Similarly, any unstable medical condition that, in the opinion of the treating physician or study investigators, would interfere with the study objectives.
6. Pregnancy or breastfeeding.
7. Major surgery within 4 weeks.
8. Concurrent use of any proton pump inhibitors, as these limit the absorption of metformin30,41.
9. History of lactic acidosis as per prior medical records or provided by the patient.
10. Metabolic acidosis, acute or chronic. Acidosis will be defined a blood pH < 7.35. Acidosis will be suspected if serum bicarbonate is < 22 mEq/L. In such cases, venous blood pH would be checked to confirm or exclude acidosis.
11. Participants with known uncontrolled diabetes, defined as a hemoglobin A1C of > 8%.
12. Participants who are already on treatment with metformin, except when metformin can be held for 4 weeks prior to the start of the study.
13. History of ongoing alcohol abuse or binge drinking. Alcohol abuse will be defined as a pattern of drinking that results in harm to one's health, interpersonal relationships, and ability to work. Binge drinking will be defined as at least one episode of consuming more than five units in men and four units in women during the previous month. One unit of alcohol can generally said to be a half pint of beer, a single measure (shot glass) of a spirit or a small glass of table wine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2016-11-15 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic Biomarker p70S6K | 28 days
  To compare the change in the pharmacodynamic biomarker p70S6K in peripheral blood T cells with the combination of metformin XR and sirolimus to that with sirolimus alone.

SECONDARY OUTCOMES:
Pharmacodynamic Biomarkers p4EBP1 and pAKT | 28 days
  To compare the changes in pharmacodynamic biomarkers p4EBP1 and pAKT in peripheral blood T cells with the combination of metformin XR and sirolimus to those with sirolimus alone.
Tolerability - Full physical Exam | 28 day cycles
  To assess the tolerability of the combination of metformin XR plus sirolimus at the selected doses a full history and physical exam will be conducted on days 1, 8, and 15.
Fasting Serum Glucose and Triglycerides | 28 days
  To compare fasting serum glucose and triglycerides on sirolimus before and after the addition of metformin XR.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Sharma, M.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States